CLINICAL TRIAL: NCT03501719
Title: Effects of ART Simplification on Inflammatory Markers in CoRis (AIR)
Acronym: AIR
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Other Study IDs: 133-17
Record Dates: First submitted 2018-03-22; First posted 2018-04-18 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: HIV
Keywords: HIV; inflammation; antiretroviral therapy; cohort studies; mortality; non-AIDS events
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Plasma samples stored at the biobank of the Spanish AIDS Research Network.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Triple ART: Patients who remain in triple ART during the follow-up.
  Interventions: Drug: Number of drugs in the ART regimen
- Dual ART: Patients switched to dual ART during the follow-up.
  Interventions: Drug: Number of drugs in the ART regimen
- Monotherapy: Patients switched to monotherapy during the follow-up.
  Interventions: Drug: Number of drugs in the ART regimen

INTERVENTIONS:
Drug: Number of drugs in the ART regimen — Triple therapy vs. dual therapy vs. monotherapy

SUMMARY:
The effects of the number of drugs included in antiretroviral therapy (ART) regimens of inflammatory markers remains undefined. We will evaluated in participants in the Spanish AIDS Research Network, whether triple ART, dual ART or monotherapy affect differentially the dynamics of inflammatory markers.

DETAILED DESCRIPTION:
During treated HIV infection, higher levels of the inflammatory and coagulation markers interleukin-6 (IL-6), D-dimers, and high-sensitivity C-reactive protein (hs-CRP) are associated with an increased risk of cardio-vascular disease (CVD), cancer, and all-cause mortality. While ART decreases IL-6, D-dimer and hs-CRP levels, these biomarkers remain elevated relative to the general population even when the plasma HIV RNA is suppressed. Markers of inflammation and coagulation have been widely studied in the general population, and related to higher risk of CVD, cancer, kidney function decline and all-cause mortality. These data collectively suggest that chronic inflammation and/or hyper-coagulation contribute to the pathogenesis of these serious non-AIDS events during otherwise effective ART. Given the assumed, albeit unproven, role of these pathways in causing disease, both vascular and non-vascular, there is intense interest in studying interventions that reduce inflammation and/or coagulation.

Recent simplification strategies have demonstrated that once HIV RNA suppression is achieved, the extent of virological control does not appear to depend so much on the number of drugs, but on the time of HIV RNA suppression before the simplification. In fact, some simplification therapies, including dual regimens based in boosted-protease inhibitors (PI) have proved to be non-inferior to triple ART, provided that drug resistance has been excluded. More recently, dual therapies based in other combinations not based in boosted-PI have emerged as viable therapeutic strategies.

While these approaches of ART simplification seems to be non-inferior to standard triple therapy in terms of short-term plasma HIV RNA suppression and CD4+ T cell count dynamics, it is unknown whether ART simplification will prove safe in the long term. Mounting evidence support that the concentration of drugs, which may be related to the number of drugs, affects the extent of virological control in the tissues in which HIV persists and replicates, generating low-level viremia and contributing to chronic inflammation. It is likely that clinical trials powered to detect differences in clinical events will not be performed. Hence, the long-term clinical efficacy of ART simplification must be assessed in cohort studies and the long-term effects on inflammatory markers that independently predict mortality must be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects initiating ART in CoRIS from 2004 with triple therapy.
* HIV RNA suppression achieved in the first 48 weeks of ART.

Exclusion Criteria:

* ART initiation with regimens with less than three drugs
* Virologic failure in the first 48 weeks of ART
* AIDS conditions or serious non-AIDS events in the first 48 weeks of ART.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Inflammation | From baseline through study completion, an average of 3 years
  Plasma IL-6 levels in plasma

SECONDARY OUTCOMES:
Immune activation | From baseline through study completion, an average of 3 years
  CD4/CD8 ratio in blood
Coagulation | From baseline through study completion, an average of 3 years
  D-dimers levels in plasma
Gut epithelial integrity | From baseline through study completion, an average of 3 years
  Intestinal fatty acid binding protein (IFABP) levels in plasma
Monocyte activation/bacterial translocation | From baseline through study completion, an average of 3 years
  Soluble CD14 levels in plasma
Immunological variables | From baseline through study completion, an average of 3 years
  Nadir CD4+ T cell count, highest CD8+ T cell count and nadir CD4/CD8 ratio.
Comorbidities | From baseline through study completion, an average of 3 years
  Number and type of comorbidities, including HCV coinfection.
Period | Baseline
  Year of ART initiation
ART history | From baseline through study completion, an average of 3 years
  Number of previous ART regimens
Available virological information | From baseline through study completion, an average of 3 years
  Number of HIV RNA determinations
ART exposure | From baseline through study completion, an average of 3 years
  Number and reasons of previous ART modifications
Sociodemographics | At baseline
  Country of origin

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided